CLINICAL TRIAL: NCT05017532
Title: Cognitive Remediation for Social Cognition in Schizophrenia and Related Disorders: Acceptability, Feasibility and Preliminary Effects of Remoted RC2S+ (RC2S+ Remote)
Brief Title: Cognitive Remediation for Social Cognition in Schizophrenia and Related Disorders
Acronym: RC2S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Martin Lepage, Clinical professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC2S
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Psychosis; Schizophrenia; Cognitive Impairment
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Intervention with RC2S+ that consists of 24 biweekly sessions
  Interventions: Behavioral: The program Remédiation Cognitive de la Cognition Sociale en Schizophrénie (RC2S+)

INTERVENTIONS:
Behavioral: The program Remédiation Cognitive de la Cognition Sociale en Schizophrénie (RC2S+) — The program Remédiation Cognitive de la Cognition Sociale en Schizophrénie (RC2S+) is a personalized CR treatment targeting social cognition (e.g. theory of mind, emotion recognition) using virtual reality to emulate daily social interactions

SUMMARY:
This study will investigate whether the remote administration of the cognitive remediation program RC2S+ acceptable and feasible in people with schizophrenia and related disorders.

DETAILED DESCRIPTION:
Schizophrenia and related psychotic disorders are associated with major functioning difficulties encompassing various areas of everyday life such as social interactions or school and work performance. Cognition, and more particularly social cognition, defined as the mental processes underlying social interactions, is considered as one of the best predictors of functioning in schizophrenia and related psychotic disorders. Social cognitive deficits thus represent a promising treatment target to promote functional recovery. Cognitive remediation (CR) is a behavioural intervention that can improve social cognitive deficits and clinical symptoms and moderate to large effect sizes have been reported. While there is great excitement that such interventions can also improve functioning, very few CR program for social cognition have used a personalized approach to tailor treatment to individual difficulties despite the benefit of personalizing CR treatment in schizophrenia. The program Remédiation Cognitive de la Cognition Sociale en Schizophrénie (RC2S+) is a personalized CR treatment targeting social cognition using virtual reality to emulate daily social interactions. Two case studies conducted in France with people with schizophrenia have demonstrated acceptability and feasibility of in-person RC2S+ while providing preliminary evidence for efficacy with the report of significant improvement of social cognitive and functional difficulties. While these preliminary results are encouraging, the program has never been used in Canada. Psychosocial intervention, and particularly those targeting social cognition, need to be culturally adapted. Thus, a preliminary study is necessary to assess if RC2S+ is culturally adapted to the social norms and rules of French and English-speaking Canadians. Further, this study needs to consider the actual context of the COVID-19 pandemic which has highlighted the important vulnerability of people with psychotic disorders and the need to adapt evidence-based interventions such as CR to increase access to mental healthcare services. Online interventions have rapidly developed in the last year in response to COVID-19 and these interventions address important factors that are known to limit access to psychiatric care in people with psychotic disorders. A remote version will however require an acceptability and feasibility assessment.

Our main objective is to assess the acceptability, feasibility, and preliminary effect of the remoted RC2S+. To reach this goal, we will, 1) Translate the RC2S+ program in English and adapt the program for French Canadians and 2) Determine the acceptability, the feasibility and the preliminary effect of the remoted RC2S+.

Twenty-six participants with a diagnosis of schizophrenia and related psychotic disorder aged 18 years or older and who present with at least one social cognitive impairment will be recruited. They will be initially assessed for social cognition as well as clinical outcomes (e.g. symptoms, recovery, functioning). Then, participants will receive 24 biweekly individual sessions of RC2S+ of 1 hour with a therapist. Intra-session questionnaires will be administered at different timepoints to the participants and the therapists to assess therapeutic alliance, motivation toward treatment as well as the satisfaction regarding treatment. At the end of treatment, participants will be reassessed with the similar measures as baseline.

This study will provide the first insight of the preliminary effect of RC2S+ administered remotely, in addition to providing French-Canadian and English version of this novel program. The results of the current study will provide relevant information to improve the program and its delivery for a future efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of schizophrenia or a related psychotic disorder
2. Being followed and treated by a clinician of the Douglas Mental Health University Hospital
3. Being 18 or older
4. Having an objective difficulty in social cognition (i.e. emotion recognition, theory of mind, attributional bias, social perception) defined as a performance equal of below 1 standard deviation from the normative group on one of the following measures: Penn Emotion Recognition Task (ER-40; Emotion recognition), Combined Stories Test (COST; Theory of mind), Social Knowledge test (SKT; Social knowledge) or Interpersonal, Personal and Situational Attributions Questionnaire (IPSAQ; Attributional style). This criterion is mandatory since we need to be able to remediate a difficulty during cognitive remediation.
5. Being considered symptomatically stable and capable of using the online platforms, as judged by their primary clinicians (i.e., psychiatrist, case manager, psychologist)
6. Having access to digital technology, Internet and access to a private space (a room where the participant can be alone)
7. Being able to nominate an emergency contact

Exclusion Criteria:

1. Evidence of an organic cause for cognitive difficulties (e.g. neurological disease, history of brain trauma)
2. History of mental retardation or autism spectrum disorder
3. Being hospitalized at the time of recruitment
4. Inability to speak or read French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Combined Stories Test (COST) | The administration time is estimated at 30 minutes.
  This test assesses Theory of Mind (ToM) abilities and includes 30 short verbal stories. Participants are asked to read each story out loud and are asked to answer ToM and control questions.
Social Knowledge Test (SKT) | The administration time is estimated at 5 minutes.
  This test assesses social knowledge. Participants are presented with a series of short hypothetical situations and are asked to state how they think most people in this situation would feel.
Penn Emotion Recognition Task (ER-40) | The administration time is estimated at 10 minutes.
  This test assesses emotion recognition on faces. A total of 40 faces are presented to the participants who must choose between five different emotions.
Interpersonal, Personal and Situational Attributions Questionnaire (IPSAQ) | The administration time is estimated at 10 minutes.
  This test assesses attributional style. Participants are presented with 32 social situations and for each of them, they must decide what was the main cause of the event described in each statement and select if the cause is whether because of them, because of another person or because of the situation.

SECONDARY OUTCOMES:
DACOBS: Davos Assessment of Cognitive Biases Scale | The administration time is estimated at 10 minutes.
  This questionnaire assesses cognitive biases through 42 items rated on a Likert scale from 1 (strongly disagree) to 7 (strongly agree).
PANSS-6: Positive and Negative Syndrome Scale | The administration time is estimated at 20 minutes.
  Through a semi-structured interview, the positive and negative symptomatology of schizophrenia is explored. In this reduced scale, the following symptoms are assessed: delusions, conceptual disorganization, hallucinations, flattened affect, passive social withdrawal, and poverty of speech.
Social Interaction Anxiety Scale (SIAS) | The administration time is estimated at 5 minutes.
  The SIAS is a 20 items self-report questionnaire to assess social anxiety. This questionnaire provides a clinical picture of the cognitive, affective, and behavioral reactions to interactional situations.
Patient Health Questionnaire (PHQ-9) | The administration time is estimated at 5 minutes.
  this questionnaire assesses the principal diagnostic criteria of major depression.
First-episode social functioning scale (FESF) | The administration time is estimated at 10 minutes.
  This self-report questionnaire aims to assess functioning in several areas including productive activities (e.g. school, work), social functioning (e.g. family, friends, acquaintances) and instrumental activities of daily living (e.g. transportation, money management). Items are rated on a Likert scale ranging from "completely disagree" to "completely agree" for the ability of the participant to perform the activity, and on a scale ranging from "Never" to "Always" for the frequency of the activity (with the option never if the activity is not performed by the participant).
The Questionnaire about the process of recovery (QPR) | The administration time is estimated at 5 minutes.
  The QPR is a 22 item self- report measure measuring the process of recovery from a psychotic disorder. The items are rated on a five-point Likert scale ranging from "strongly disagree" to "strongly agree".

OTHER OUTCOMES:
NIMH suicide screening questionnaire (NIMH-SSQ) | The administration time is estimated at 5 minutes.
  This questionnaire includes five questions to screen for suicide risk.
Échelle de repercussions fonctionnelles des troubles de la cognition sociale (ERF-CS) | The administration time is estimated at 10 minutes.
  This short semi-structured interview explores the presence and impact of various social cognitive deficits in everyday life. The interview also assesses how much the participant is bothered by these difficulties.
Goal Attainment Scale (GAS) | The administration time is estimated at 5 minutes.
  The GAS is a flexible scale that allows the elaboration of personalized objectives before starting treatment that will be reassessed at follow-ups. The scale is rated on a scale from -2 to +2. A score of 0 indicates that the participant has reached his initial goal. Scores of +1 or +2 are obtained if the participant has exceeded or greatly exceeded his initial goal. Scores of -1 and -2 are obtained if the participant did not completely or not all reached his objective. When the objectives are set, an operational definition is established for each level of ratings.
MUSIC® Model of Motivation Inventory, Cognitive Training version (MMI-CT) | The administration time is estimated at 5 minutes.
  The MMI-CT is an 18-item self-report questionnaire that assesses motivation toward cognitive training. The questionnaire is divided into five scales namely empowerment, usefulness, success, interest and caring. Responses range from 1 (Strongly disagree) to 6 (Strongly Agree).
Working Alliance Inventory Short form (WAI) | The administration time is estimated at 5 minutes.
  The WAI I is a self-report questionnaire of 36 items rated on a Likert scale from 1 (Never) to 7 (Always) to assess therapeutic alliance.
eTherapy Attitudes and Process questionnaire (eTAP) | The administration time is estimated at 5 minutes.
  The eTAP is a self-report questionnaire that measures factors related to client engagement in e-interventions for mental health. There are 16 questions rated on a Likert scale ranging from 1 to 7.
RC2S+ Acceptability, Usability, Safety, Impact, and Satisfaction Questionnaire (RC2S+-AUSIS-Q) | The administration time is estimated at 5 minutes.
  This questionnaire was built for this project, based on a similar questionnaire created by our team in a previous project (iCog-AUSI-Q).

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thibaudeau E, Peyroux E, Franck N, Carling H, Lepage M. Navigating Social Cognitive Impairments in Schizophrenia Spectrum Disorders: Protocol for a Pilot Pre-Post Quasi-Experimental Study for Remote Avatar-Assisted Cognitive Remediation Therapy. JMIR Res Protoc. 2024 Mar 13;13:e54251. doi: 10.2196/54251. PMID 38477975